CLINICAL TRIAL: NCT00650182
Title: Safety Evaluation of D-TRANS Fentanyl With Naltrexone HCL in Opioid Tolerant Patients (ALZA C-2002-022)
Brief Title: A Study to Evaluate the Safety of D-TRANS Fentanyl With Naltrexone in Adult Patients With Chronic Pain and Who Are Opioid Tolerant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006715
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Chronic Pain
Keywords: patch; fentanyl; chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Fentanyl; Naltrexone

INTERVENTIONS:
Drug: fentanyl; naltrexone

SUMMARY:
The primary objective was to evaluate the safety of D-TRANS fentanyl with naltrexone HCl system compared to the Duragesic (fentanyl transdermal system) in opioid tolerant patients.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, double-dummy safety study in adult patients who required continuous opioid treatment for chronic pain. Patients had to be on a stable dose of duragesic for 21 days prior to the start of the study treatment period and have completed a screening period of at least 14 days to enter this study. Eligible patients were randomized (2:1) to receive the equivalent strength of D-TRANS fentanyl with naltrexone HCl (and placebo Duragesic) or the same dose of Duragesic (and placebo D-TRANS fentanyl with naltrexone HCl [D-TRANS fentanyl with naltrexone]) for a 15-day treatment period. If necessary, patients could be titrated to higher or lower doses during the 15-day treatment period. Each system was worn for 72 hours then replaced by a new system until the end of the 15-day treatment period. Patients were telephoned 3 times a day during the first 3 days of the study and then once daily for the remainder of the study to determine if there were any signs of opiate overdose or withdrawal. The patient was to be followed as medically indicated based on the responses to the questions. Safety assessments included summarizing the incidences of adverse events (including topical adverse events), vital signs measurements, and clinical laboratory evaluations. Blood samples were also collected for analysis of naltrexone and fentanyl concentrations at scheduled times during the study. Efficacy assessments included patient global assessments, investigator global assessments, pain intensity, and brief pain inventory. Blood samples were also to be collected for analysis of naltrexone and fentanyl prior to any dose change and if a patient experienced a serious adverse event possibly or probably related to study drug. Duragesic delivering fentanyl doses of 25 mcg/h, 50 mcg/h, 75 mcg/h, or 100 mcg/h, and a D-TRANS placebo on Days 1, 4, 7, 10, and 13 or D-TRANS fentanyl with naltrexone delivering fentanyl doses of 25 mcg/h, 50 mcg/h, 75 mcg/h, or 100 mcg/h, and a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pain who require continuous opioid analgesia
* Must enter the study on a stable dose of Duragesic for at least 21 days and consent to use a medically acceptable method of contraception throughout the entire study, and for females 1 week after the study is completed and for males 3 months after the study is completed.

Exclusion Criteria:

* Skin disease that precluded the use of a transdermal system
* Clinically significant laboratory abnormalities
* Significant mental status changes that result in disorientation, memory impairment, or inability to report accurately
* Illicit drug, prescription drug, or alcohol abuse
* Cardiopulmonary disease
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2003-01; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety of 2 transdermal formulations of fentanyl (D-TRANS fentanyl with naltrexone transdermal system and Duragesic (fentanyl transdermal system) in patients with chronic pain who were opioid tolerant.

SECONDARY OUTCOMES:
Efficacy assessments included patient global assessments, investigator global assessments, pain intensity, and brief pain inventory. Blood samples were also to be collected for analysis of naltrexone and fentanyl prior to any dose change.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- See also: Click here to view the journal abstract from the study manuscript. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=107&filename=CR006715_CSR.pdf